CLINICAL TRIAL: NCT01659177
Title: The Effect of Food on the Pharmacokinetics of LY2140023 and LY404039 in Healthy Subjects After Administration of the Commercial Tablet Formulation of LY2140023
Brief Title: A Study of LY2140023 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to stop the trial was based on efficacy results in the overall schizophrenia patient population.
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14511; H8Y-MC-HBDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2012-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — LY 2140023

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2140023 fasting (Experimental): Single oral dose of 80 mg LY2140023 given in fasted state
  Interventions: Drug: LY2140023
- LY2140023 + food (Experimental): Single oral dose of 80 mg LY2140023 given after standardized high-fat breakfast
  Interventions: Drug: LY2140023

INTERVENTIONS:
Drug: LY2140023 — Administered orally

SUMMARY:
The study will evaluate the effect of food on absorption of LY2140023 in blood. This study involves a single dose of 80 mg LY2140023 taken as a tablet by mouth on 2 occasions, once on an empty stomach and once after eating breakfast. There is a minimum 3 day washout between doses. This study will last approximately 16 days not including screening. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males or females, as determined by medical history and physical examination
* Male participants agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023, and agree not to donate sperm for 3 months following the last dose of LY2140023
* Female participants:

  * of childbearing potential, who test negative for pregnancy at screening and who agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023
  * of non-childbearing potential i.e. postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy or confirmed tubal occlusion (not tubal ligation). Postmenopausal is defined as spontaneous amenorrhea for at least 12 months, and a plasma follicle-stimulating hormone (FSH) level >40 milli-international units per milliliter (mIU/mL), unless the participant is taking hormone replacement therapy
  * have given written informed consent approved by Lilly and the chosen ethical review board (ERB)

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 90 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2140023 or LY404039, related compounds, activated charcoal, or any components of the formulation
* Are persons who have previously withdrawn from this study or any other study investigating LY2140023 after receiving at least 1 dose of LY2140023
* Show evidence or any history of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* Have increased risk of seizures based on a history of:

  * one or more seizures (except for a single simple febrile seizure [lacking focality and lasting less than 15 minutes, not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * head trauma with loss of consciousness or a post-concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * CNS infection, uncontrolled migraine or transient ischemic attack (TIA) within 1 year; stroke with persistent neurological deficit (focal or diffuse), uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning. TIA is defined as "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * brain surgery
  * electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, or sharp-slow wave complexes, or as locally defined)
  * brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (except hydrocephalus treated by shunt and without neurological deficit)
* Show evidence of active renal disease (for example, diabetic renal disease, polycystic kidney disease) or creatinine clearance less than 90 milliliters per minute (mL/min) as determined by the Cockroft Gault formula
* Show evidence or any history of known substance dependence or abuse at any time (according to Diagnostic and Statistical Manual of Mental Disorders [DSM-IV] diagnosis), or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a clinically significant abnormality in the neurological examination
* Participants judged prior to randomization to be at suicidal risk by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum concentration (Cmax) of LY2140023 and LY404039 | Up to 24 hours after administration of study drug
Pharmacokinetics: Area under the concentration curve (AUC) of LY2140023 and LY404039 | Up to 24 hours after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allschwil, Switzerland